CLINICAL TRIAL: NCT02728661
Title: Patient-Centered Weight Loss Program for Knee Replacement Patients
Acronym: PACE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K12HS023011 (AHRQ)
Record Dates: First submitted 2016-03-29; First posted 2016-04-05 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: ARTHROPLASTY, REPLACEMENT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PACE (Experimental): PACE participants will begin up to 6 weeks prior to their scheduled TKR and continue until 12 weeks after their TKR. Participants will be given personalized weight, dietary, and physical activity goals. Participants will be encouraged to monitor their dietary intake and physical activity using their preferred method of self-monitoring. Participants will have regular contact with their coaches either in-person or over the telephone on a weekly or bi-weekly basis, based on preference during the first 14 weeks (from up to 6 weeks pre-op to 12 weeks post-op). Further, participants may opt to receive regular text messages or emails from coaches if they prefer. At 12 weeks, PACE participants will enter a maintenance period and not have any contact with coaches.
  Interventions: Behavioral: PACE
- Delayed PACE (Experimental): After being notified of their randomized condition at baseline (up to 6 weeks prior to surgery), Delayed PACE participants will not have contact with coaches until 12 weeks after surgery. At 12 weeks after surgery, Delayed PACE participants will be given personalized weight, dietary, and physical activity goals. Participants will be encouraged to monitor their dietary intake and physical activity using their preferred method of self-monitoring. Participants will have regular contact with their coaches either in-person or over the telephone on a weekly or bi-weekly basis, based on preference during the first 14 weeks. Further, participants may opt to receive regular text messages or emails from coaches if they prefer.
  Interventions: Behavioral: Delayed PACE

INTERVENTIONS:
Behavioral: PACE — PACE is an 14 week behavioral weight loss intervention developed specifically for knee replacement patients that starts up to 6 weeks prior to surgery.
  Arms: PACE
Behavioral: Delayed PACE — Delayed PACE is an 14 week behavioral weight loss intervention developed specifically for knee replacement patients that starts 12 weeks after surgery.
  Arms: Delayed PACE

SUMMARY:
PACE is a patient-centered weight loss program that was developed specifically for knee replacements based on input from stakeholders, including knee replacement patients, physical therapists, and orthopedic surgeons. In this pilot study, participants undergoing knee replacement will be randomized to either start a weight loss program before surgery (PACE) or after surgery (Delayed PACE). Both programs will receive a 14-week intervention and complete assessments at baseline (up to 6 weeks prior to surgery), 12 weeks after surgery, and 26 weeks after surgery.

DETAILED DESCRIPTION:
It is estimated that half of patients diagnosed with knee osteoarthritis (OA) will need a total knee replacement (TKR) during their lifetime. Of patients who need a TKR, 80-95% are overweight or obese. While patients are encouraged to lose weight, limited, if any, guidance is provided to achieve recommended weight loss. Many patients perceive that TKR is a necessary precursor for the initiation of weight loss. Yet, 66% of patients actually gain weight by 2 years after surgery. Patients undergoing TKR not only face unique barriers (i.e., pain, mobility limitations, motivation) to weight loss, but also have to balance pre- and post-operative concerns from physicians, surgeons, and rehabilitation specialists. To best accommodate the needs of both patients (pre- and post-TKR) and healthcare professionals (i.e., surgeon, physical therapist), patient and stakeholder engagement and activation is imperative in the development of a patient-centered weight loss intervention. Investigators completed 20 interviews with patients pre- and post-TKR and identified weight loss barriers, preferred intervention components (e.g., delivery method, contact frequency, self-monitoring modality) and patient-reported outcomes (e.g., physical function, pain) viewed as critical by patients. Investigators developed a patient-centered weight loss program (PACE) guided by these results and additional input from stakeholders to meet the needs of patients and healthcare professionals. PACE is a randomized pilot study comparing weight loss and patient-reported outcomes between PACE (program starting up to 6 weeks pre-TKR to 12 weeks post-TKR) and Delayed PACE (program starting 12 weeks post-TKR to 26 weeks post-TKR).

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25-45 kg/m2
* Have a scheduled knee replacement at least 1 week away from baseline assessment
* Obtain physician approval to participate
* English speaking
* willing to attend 3 in-person assessments.

Exclusion Criteria:

* Have any contraindications to diet or weight loss
* Undergoing simultaneous bilateral knee replacement or have a scheduled or anticipated knee replacement for the contralateral knee in the next 26 weeks
* Have a mobility limiting comorbidity besides relating to TKR
* Taking anti-obesity medications
* Enrolled in a formal weight loss program
* Have had or is planning to have bariatric/gastric/lapband surgery
* Is planning to relocate out of the Chicago land area in the next 12 months.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-05; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in weight measured with a balance-beam scale | Change from baseline to 12 and 26 weeks

SECONDARY OUTCOMES:
Change in physical function assessed by the timed up and go | Change from baseline to 12 and 26 weeks
Change in pain measured by WOMAC | Change from baseline to 12 and 26 weeks

OTHER OUTCOMES:
Change in physical activity objectively-measured with accelerometry | Change from baseline to 12 and 26 weeks
Behavioral adherence assessed by session and self-monitoring completion | 26 weeks post-op

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PACE Research Study — https://sites.northwestern.edu/pacestudy/info/